CLINICAL TRIAL: NCT03935581
Title: Assessment of Safety and Feasibility of ExAblate Neuro System to Perform Auto-Focusing Echo Imaging in Patients With Idiopathic Essential Tremor With Medication Refractory Tremor
Brief Title: Safety and Feasibility of ExAblate Neuro System to Perform Auto-Focusing Echo Imaging in Patients With Essential Tremor
Acronym: ET004
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: InSightec (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: ET004
Record Dates: First submitted 2019-04-18; First posted 2019-05-02 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Tremor, Essential; Neurologic Manifestations; Tremor
Keywords: MRgFUS; ExAblate; Essential Tremor; Auto-Focusing Echo Imaging
MeSH Terms: conditions — Essential Tremor; Neurologic Manifestations; Tremor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ExAblate 4000 System (Experimental): ExAblate Neuro system to perform AF echo imaging in treatment of Essential Tremor
  Interventions: Device: ExAblate

INTERVENTIONS:
Device: ExAblate — Auto Focusing (AF) echo imaging

SUMMARY:
The objective of this study is to evaluate the safety and feasibility of Auto Focusing (AF) echo imaging using the ExAblate Neuro system

DETAILED DESCRIPTION:
This clinical investigation is a feasibility study designed to evaluate the safety and feasibility of the ExAblate Neuro system to perform AF echo imaging in patients diagnosed with idiopathic Essential Tremor. during the standard care procedure for ET, patients will be injected with Definity microbubbles which will enable the ExAblate Neuro system to perform the AF imaging.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female age 22 years or older
2. Able and willing to give consent and able to attend all study visits
3. A confirmed diagnosis of Essential Tremor resistant to medication therapy
4. Able to fit into MRI unit
5. Able to tolerate the procedure with or without some form of sedation
6. Able to communicate sensations during the ExAblate MRgFUS procedure
7. Able to activate Stop Sonication button during the ExAblate MRgFUS procedure

Exclusion Criteria:

1. Presence of unknown or MRI unsafe devices anywhere in the body.
2. Patients with known intolerance or allergies to the MRI contrast agents
3. Women who are pregnant
4. Patients with advanced kidney disease or on dialysis
5. Significant cardiac disease or unstable hemodynamic status
6. Patients exhibiting any behavior(s) consistent with ethanol or substance abuse
7. History of a bleeding disorder
8. Patients receiving anticoagulant or drugs known to increase risk of hemorrhage
9. Patients with cerebrovascular disease
10. Patients with brain tumors
11. Individuals who are not able or unwilling to tolerate the required prolonged stationary position during treatment (approximately 2-3 hours)
12. Patients who are currently participating in another clinical investigation
13. Patients unable to communicate with the investigator and staff
14. Patients who have cardiac shunts
15. Patients with relative contraindications to Definity ultrasound contrast agent including subjects with a family or personal history of arrhythmia's
16. Patients with chronic pulmonary disorders
17. Patients with a history of drug allergies, uncontrolled asthma or hay fever
18. Patients who have had deep brain stimulation or a prior neuroablative procedure
19. Women who are pregnant or nursing
20. Patients who have been administered botulinum toxins into the arm, neck, or face for 5 months prior to enrollment in the study.

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-04-25 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Device and Procedure related Adverse Events | Treatment through 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Nir Lipsman, Principal Investigator — Sunnybrook Health Science Centre
Locations (2):
- Sunnybrook, Toronto, Ontario, Canada
- Yonsei University Health System, Severance Hospital, Seoul, Seodaemun-gu, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chang KW, Rachmilevitch I, Chang WS, Jung HH, Zadicario E, Prus O, Chang JW. Safety and Efficacy of Magnetic Resonance-Guided Focused Ultrasound Surgery With Autofocusing Echo Imaging. Front Neurosci. 2021 Jan 12;14:592763. doi: 10.3389/fnins.2020.592763. eCollection 2020. PMID 33510610
- [Derived] Jones RM, Huang Y, Meng Y, Scantlebury N, Schwartz ML, Lipsman N, Hynynen K. Echo-Focusing in Transcranial Focused Ultrasound Thalamotomy for Essential Tremor: A Feasibility Study. Mov Disord. 2020 Dec;35(12):2327-2333. doi: 10.1002/mds.28226. Epub 2020 Aug 20. PMID 32815611